CLINICAL TRIAL: NCT03520894
Title: Radiotherapy in Preoperative Setting With CyberKnife as Treatment in Early Breast Cancer: an Explorative Study
Brief Title: Radiotherapy in Preoperative Setting With CyberKnife for Breast Cancer
Acronym: ROCK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Full Professor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROCK
Record Dates: First submitted 2018-04-19; First posted 2018-05-11 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant radiotherapy arm (Experimental): Early breast cancer patients eligible for breast conservative surgery will undergo neoadjuvant radiotherapy with Cyberknife robotic system
  Interventions: Radiation: Neoadjuvant radiotherapy

INTERVENTIONS:
Radiation: Neoadjuvant radiotherapy — single 21 Gy fraction of Radiotherapy before surgery

SUMMARY:
The aim of this study is to prospectively evaluate, in patients affected by early breast cancer, safety and feasibility of single fraction radiotherapy with Cyberknife R in preoperative setting, and to identify factors predictive for outcome based on biologic and clinical parameters.

DETAILED DESCRIPTION:
Monocentric, open-label, single-arm phase II study evaluating safety and efficacy of neoadjuvant radiotherapy in early breast cancer patients. Patients eligible are women aged 50 or more years old, affected by histologically proven invasive breast cancer, with positive hormonal receptors, grading 1 or 2, HER-2 negative, without lymphovascular invasion, and tumour size up to 2 cm (measured on mammography, ultrasound or magnetic resonance), negative clinical nodal status, eligible for BCS.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Women ≥ 50 years old
3. Histological diagnosis of invasive breast cancer
4. ER positive (≥ 10% of tumoral cells present ER) and/or PR positive (≥ 10% of tumoral cells present PR)
5. Grading 1 or 2
6. Her2 negative (IHC 0-1+; in patients with IHC 2+, absence of amplification at FISH
7. No lymphovascular invasion evidence at biopsy
8. Early breast cancer (T1 N0 M0) clinically and radiologically defined (ultrasound study/ magnetic resonance)
9. Patients eligible for BCS.

Exclusion Criteria:

Extension of breast disease within 5 mm from the skin surface 2. Tumor size > 2 cm 3. Patients affected by collagenopathies 4. Patients with BRCA1/2 mutations 5. Previous irradiation to homolateral breast 6. Previous irradiation to homolateral thoracic wall 7. DCIS and/or Paget's disease 8. Psychiatric disorders preventing informed consent signature.

-

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 25 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of acute skin toxicity events, measured according to RTOG/EORTC scale | 15 days
  Acute skin toxicity (from the end of radiotherapy to surgery) according to Radiation Therapy Oncology Group (RTOG)/ European Organization for research and treatment of cancer (EORTC) scale. Measuring acute skin toxicity from a minimum of 0 (no change over baseline) to a maximum of 4 (Ulceration, Hemorrage, necrosis)

SECONDARY OUTCOMES:
Number of patients with pathologic complete response (pCR) after surgery,according to Chevalier score | 30 days
  Rate of pCR according to Chevalier score
Number of patients with complete resection after surgical excision | 30 days
  Rate of complete resection R0 with margin<1cm (except for deep margin)
Number of patients free from locoregional progression at 36 months | 36 months
  locoregional progression free survival measured at 36 months
Number of patients free from metastatic progression at 36 months | 36 months
  Metastasis progression free survival measured at 36 months
Number of patients dying for breast cancer at 36 months | 36 months
  cause-specific free survival measured at 36 months
Number of patients dying for any cause at 36 months | 36 months
  global survival measured at 36 months
Rate of chronic skin toxicity events, measured according to CTCAE | 90 days
  Incidence of chronic skin toxicity (over 90 days since the end of radiotherapy; fibrosis, telangiectasia, tardive oedema) according to Common terminology criteria for adverse events (CTCAE) v 4.03. From a minimum of 1 (Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated
  * to a maximum of 4 (Life-threatening consequences; urgent intervention indicated
Rate of chronic extra-cutaneous toxicity, measured according to CTCAE | 90 days
  Incidence of chronic extra-skin toxicity (over 90 days from the end of radiotherapy; lung fibrosis, pericarditis, myocardial ischemia, valvulopathy, thoracic wall pain, fracture) according to according to Common terminology criteria for adverse events (CTCAE) v 4.03. From a minimum of 1 (Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated
  * to a maximum of 4 (Life-threatening consequences; urgent intervention indicated
Correlation of differential genetic expression, immunologic and histopathologic features of tumor sample and biomarkers in blood and urine samples with toxicity and rate of response to radiotheraèy | 60 days
  Radiogenomic: confirm of differential genetic expression of genes already validated in previous literature (30-Radiation- induced gene signature; AOI 16-gene breast signature; IRDS gene signature) with Next Generation Sequencing (NGS, RNA-seq) or Real Time PCR on frozen biopsy tissue.
  Immunologic: quantitative analysis of infiltrating leucocytes (MS and M1 macrophages, CD8+ and CD4+ lymphocytes) with immunohistochemistry on fresh biopsy tissue Histopathologic: qualitative analyses (pericytes) and quantitative pattern of vascularization in immunohistochemistry.
  Biochemical: analysis of oxidative stress markers on peripheral blood and urines:
  a) 1 hour before SBRT; b) 1 hour after SBRT; c) 1 week after SBRT; d) during 24 hours before BCS; e) during 2-4 weeks after BCS.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Livi, Prof, Study Chair — AOU Careggi; Icro Meattini, Prof, Study Chair — AOU Careggi; Giulio Francolini, MD, Principal Investigator — AOU Careggi; Vanessa Di Cataldo, MD, Principal Investigator — AOU Careggi
Locations (1):
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meattini I, Guenzi M, Fozza A, Vidali C, Rovea P, Meacci F, Livi L. Overview on cardiac, pulmonary and cutaneous toxicity in patients treated with adjuvant radiotherapy for breast cancer. Breast Cancer. 2017 Jan;24(1):52-62. doi: 10.1007/s12282-016-0694-3. Epub 2016 Mar 30. PMID 27025498
- [Background] Livi L, Meattini I, Marrazzo L, Simontacchi G, Pallotta S, Saieva C, Paiar F, Scotti V, De Luca Cardillo C, Bastiani P, Orzalesi L, Casella D, Sanchez L, Nori J, Fambrini M, Bianchi S. Accelerated partial breast irradiation using intensity-modulated radiotherapy versus whole breast irradiation: 5-year survival analysis of a phase 3 randomised controlled trial. Eur J Cancer. 2015 Mar;51(4):451-463. doi: 10.1016/j.ejca.2014.12.013. Epub 2015 Jan 17. PMID 25605582